CLINICAL TRIAL: NCT07088822
Title: A Phase 1 Study Evaluating the Safety, Tolerability, and Immunogenicity of V4020 Vaccine in Healthy Volunteers
Acronym: VEEV
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medigen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: USUHS.2025-145
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Venezuelan Equine Encephalitis; Venezuelan Equine Encephalitis Virus Infection
Keywords: VEE; VEEV; Venezuelan equine encephalitis; Live attenuated vaccine; Biowarfare; Biodefense
MeSH Terms: conditions — Encephalomyelitis, Venezuelan Equine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment This study is a Phase 1, randomized, double-blind, placebo-controlled, escalating, single-center study to evaluate the safety and immunogenicity of the V4020 vaccine in a two dose series at days 0 and 56. A second dose will be given on day 56 via the same route of administration as on day 0, but will only be administered to participants not developing a plaque-reduction neutralization assay titer (PRNT80) against V4020 of >1:20 by day 28. This will include those in the placebo-only groups. There will be three escalating dose groups of 13 participants each for 39 healthy male and healthy non-pregnant female participants 18-50 years old.
Who Masked: Participant, Care Provider, Investigator
Masking Description: During the randomized phase, Sponsor personnel and the site pharmacist will be unblinded while the investigator, clinical site, and participants participating in the study will remain blinded.
  The study is designed to keep participants and investigators blinded until completion of the clinical phase of the trial and monitoring of the clinical data. During the study all efforts will be made to keep participants and investigators unaware of participant assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Group 1 will receive an administration on day 0 (and possibly also day 56) of Subcutaneous route of dose escalation.
  1. Low dose: A single dose of plaque forming units (PFU) administered 10^4 subcutaneously.
  2. Medium dose: A single dose of 10^5 PFU administered subcutaneously.
  3. High dose: A single dose of 10^6 PFU administered subcutaneously
  Interventions: Biological: V4020
- Group 2 (Experimental): Group 2 will receive an administration on day 0 (and possibly also day 56) of Intramuscular route of dose escalation.
  1. Low dose: A single dose of plaque forming units (PFU) administered 10^3 PFU intramuscularly.
  2. Medium dose: A single dose of 10^4 PFU intramuscularly.
  3. High dose: A single dose 10^5 PFU intramuscularly.
  Interventions: Biological: V4020
- Group 3 (Experimental): Group 3 will receive an administration on day 0 (and possibly also day 56) of placebo (10:3 allocation).
  Interventions: Biological: V4020

INTERVENTIONS:
Biological: V4020 — The V4020 vaccine was prepared using an iDNA® infectious clone that encodes the full-length rearranged genomic RNA downstream from the optimized CMV promoter. Compared to the wild type VEEV, V4020 contains genetic rearrangement within the genomic RNA, with the capsid gene placed downstream from the glycoprotein genes. V4020 also includes attenuating mutations from the VEE TC83 vaccine, nucleotide A at position 3 in the untranslated region and E2-120Arg in the E2 glycoprotein. Notably, the E2-120Arg attenuating mutation was genetically engineered in V4020 to prevent reversion mutations. The E2-120Arg was encoded in V4020 by a CGA codon instead of AGA in the TC83 virus. Therefore, in the V4020 vaccine, at least two mutations would be needed to revert to the wildtype ACA (E2-120Thr). In contrast, in the TC83 vaccine, an AGA codon encodes the attenuating mutation E2-120Arg, and a single point mutation would be sufficient to revert to the 213 VEEV wild type ACA (E2-120Thr).

SUMMARY:
The purpose of the study is to evaluate the safety and immunogenicity of a novel Venezuelan Equine Encephalitis virus (VEEV) vaccine (V4020) for the first time in humans compared to placebo when administered by subcutaneous or intramuscular injection.

DETAILED DESCRIPTION:
The primary objective of the study will be to measure safety. The primary endpoint measures to assess this objective will include but not be limited to

* Frequency and nature of adverse events (AEs) reported or observed in participants;
* Relatedness between AEs and vaccine administration;
* Interventions or therapy required by participants experience vaccine related adverse events;
* Resolution or outcome of AEs. Secondary Objectives and Endpoints Two main immunogenicity objectives will be assessed to include the number considered adequately immunized, and the magnitude and durability of titer responses.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all the following criteria to be included in the study:

  1. 18-50 years old at time of consent.
  2. Have VEE virus PRNT80 < 1:10.
  3. If biologic female of childbearing potential, must agree to have a serum pregnancy test 3 days before vaccine administration. (Exceptions for those with documented hysterectomy or ≥ 3 years of menopause.) The results must be negative. Females of child-bearing potential must agree not to become pregnant for at least 3 months after receipt of vaccination. They must also agree to use an acceptable form of birth control with less than a 1% failure rate as determined by the US Centers for Disease Control (https://www.cdc.gov/reproductivehealth/ contraception/index.htm).
  4. Sign and date the approved informed consent document, a separate consent form for HIV testing, and HIPAA Authorization.
  5. Medical exam (including history, concomitant medications, physical examination, and laboratory tests) negative for acute morbidities within 60 days of planned first administration of vaccine.
  6. Be willing to return for all follow-up visits.
  7. Maintain a symptom diary and bring it to all follow-up appointments. Participants will be provided a template and instructed on how to record dates, times, and details of relevant symptoms (e.g. severity, concurrent activity).
  8. Agree to report any AEs that may or may not be associated with administration of the vaccine for at least 28 days after administration and agree to report all SAEs (for example, resulting in hospitalization) for the duration of participation in the study.
  9. Agree to take appropriate measures to avoid mosquito and other insect bites if experiencing vaccine-related symptoms following vaccination until those symptoms resolve, and/or tests for vaccine virus shedding become negative.
  10. Agree to defer blood, bone marrow and organ donation for 1 year after vaccine receipt.

Exclusion Criteria:

* Participants meeting any of the following criteria will be excluded from the study:

  1. Have received experimental VEE vaccine previously or had known VEE exposure.
  2. Have family history (first degree relative) of diabetes mellitus (any type), a personal or family history of gestational diabetes, a confirmed elevated fasting serum glucose test (> 125 mg/dL), or a hemoglobin A1c > 5.6%. (At the PI's discretion, a participant may enroll if the family history of diabetes is only of late onset in an elderly parent.)
  3. Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical examination, EKG, and/or laboratory screening test.
  4. Have a personal history of an immunodeficiency or received treatment with an immunosuppressive medication, such as systemically administered glucocorticoids (e.g., prednisone) within

  <!-- -->

  1. month before planned administration of the vaccine or with other immunosuppressive therapies within 6 months of planned administration of the vaccine. Other immunosuppressive therapies include all cancer chemotherapeutic agents, drugs to prevent transplant rejection, interferons, monoclonal antibodies, protein kinase inhibitors, methotrexate, TNF (tumor necrosis factor) inhibitors, and any other clinically significant immunosuppressive medication as determined by the PI. Current administration of topical, inhalational, or intranasal glucocorticoids is not excluded. 5. Breastfeeding female. 6. Have any known allergies to components of the vaccine. 7. Receipt or planned receipt of any experimental or licensed vaccine, except for a licensed seasonal influenza, coronavirus, or other required health maintenance vaccine, within the period 30 days prior to initial injection through 60 days after the Day 70 follow-up. (~ 6-month period in total) 8. A history of prior vaccination against or confirmed infection with eastern equine encephalitis (EEE) virus, western equine encephalitis (WEE) virus, chikungunya (CHIK) virus or Venezuelan equine encephalitis (VEE) Virus. Those found to have pre-existing protective antibody responses against VEEV at baseline will also be excluded. 9. Have any unresolved AE resulting from a previous immunization. 10.Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child. 11. Syncopal episode within 12 months of screening. 12.Suspected or known current alcohol abuse as defined by the American Psychiatric Association in DSM V (Diagnostic and Statistical Manual of Mental Disorders-5th edition) 13.Chronic or active illicit and/or intravenous drug use by history. 14.Any other significant finding that, in the opinion of the investigator, would increase the risk of the individual having an adverse outcome from participating in this study. 15.Have an acute or chronic medical condition that, in the judgment of the PI, would impact participant safety. 16.Have been in contact with a suspected COVID-19, influenza and/or RSV patient within the past 14 days will need to wait an additional 14 days or have negative test laboratory test results before enrolling. 17.Participants who are likely to have direct contact with all equine species (e.g., equestrians, horse farmers) during the clinical trial period will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety | 28 days
  Primary Outcome Measure:
  1. Primary Outcome Measures
  •Percentage of participants for each study group and overall reporting 1 or more unsolicited Adverse Events (AEs) of probable or definite relatedness by severity grade using the current version of the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials Criteria for Adverse Events (CTCAE). Primary safety endpoints will be based on solicited adverse events during the first 28 days postvaccination following each vaccination. Serious adverse events will be solicited and reported throughout the trial. •Percentage of participants for each study group and overall reporting systemic vaccine reactogenicity by severity, and association with vaccination based on a diary and clinical evaluation. Reactogenicity will be reviewed using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in preventative Vaccine Clinical Trials FDA Guidance, September 2007.

CONTACTS AND LOCATIONS:
Locations (1):
- Uniformed Services University of the Health Sciences, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32121666/